CLINICAL TRIAL: NCT06443697
Title: A Machine Learning-based Prediction Model for Delayed Clinically Important Postoperative Nausea and Vomiting in High-risk Patients Undergoing Laparoscopic Gastrointestinal Surgery
Brief Title: A Machine Learning Prediction Model for Delayed CIPONV
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhi-Nan Zheng, Attending doctor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2024ZSLYEC-202
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delayed CIPONV: Patients experiencing CIPONV between 25 and 120 hours post-surgery.
  Interventions: Other: No intervention
- Non-delayed CIPONV: Patients not experiencing CIPONV between 25 and 120 hours after surgery.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a secondary analysis and no intervention is implemented.

SUMMARY:
Postoperative nausea and vomiting (PONV) can lead to serious postoperative complications, but most symptoms are mild. Clinically important PONV (CIPONV) refers to PONV symptoms that have a significant impact on the patient's well-being and recovery. Present predictive systems for PONV are mainly concentrated on early PONV. However, there is currently no suitable prediction model for delayed PONV, particularly delayed CI-PONV. This study aims to develop and validate a prediction model for delayed CI-PONV using machine learning algorithms utilizing perioperative data from patients undergoing laparoscopic gastrointestinal surgery.

All 1154 patients in the FDP-PONV trial will be enrolled in this study. Delayed CIPONV is defined as experiencing CIPONV between 25-120 hours after surgery. After selecting the modeling variables from 81 perioperative clinical features, six machine learning models are established to generate the risk prediction models for delayed CIPONV. The area under the receiver operating characteristic curve, accuracy, sensitivity, specificity, positive predictive value, negative predictive value, F1 score and Brier score are used to evaluate the model performance. Shape Additive explanation analysis was conducted to evaluate feature importance.

DETAILED DESCRIPTION:
The website https://mvansmeden.shinyapps.io/BeyondEPV/ was used for sample size calculation, considering 6 candidate predictors, an event fraction of 0.14, and a criterion value for reduced mean predictive squared error of 0.03. The calculated sample size is 1080, with a minimally required expected event per variable of 25.1. Therefore, a sample size of 1154 patients is deemed sufficient to support the inclusion of 6 predictors in the development of the predictive model.

A total of 81 variables, including demographics, comorbidities, laboratory findings, as well as information related to anesthesia and surgery, are prospectively collected in the FDP-PONV trial and considered as potential predictive factors in this study. The least absolute shrinkage and selection operator method is used to identify clinically significant variables. Further selection of the final predictors is performed using stepwise regression based on the Akaike Information Criterion.

The entire dataset is randomly divided into a training set and a validation set in a ratio of 7:3. Six machine learning models, namely logistic regression, random, extreme gradient boosting, k-nearest neighbor, gradient boosting decision, and multi-layer perceptron, were developed to create risk prediction models for delayed CIPONV. The performance of the models is assessed by comparing the area under the receiver operating characteristic curve, accuracy, sensitivity, specificity, positive predictive value, negative predictive value, F1 score, Brier score and calibration curve. Bootstrap resamples is conducted 1000 times on the training cohort to evaluate the predictive model's performance. Decision curve analysis is conducted to assess the clinical applicability of the model. The SHapley Additive Explanations library (SHAP) is used to interpret the prediction model.

ELIGIBILITY:
Inclusion Criteria:

a) age between 18 and 75 years, b) having 3 or 4 Apfel risk factors, and c) scheduled to undergo laparoscopic gastrointestinal surgical procedures under general anesthesia.

Exclusion Criteria:

a) American Society of Anesthesiologists (ASA) physical status greater than 3, b) severe hepatic dysfunction, c) contraindications to fosaprepitant, 5-HT3 receptor antagonist, or dexamethasone, d) preoperative use of medications known to have antiemetic properties, e) presence of mental disorders or inability to communicate, and f) pregnant or nursing women.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All 1154 patients in the FDP-PONV trial will be enrolled in this study. The FDP-PONV trial was a randomized, controlled, double-blind trial that aimed to evaluate the effectiveness and safety of fosaprepitant in managing PONV in patients undergoing laparoscopic gastrointestinal surgery. The FDP-PONV trial was approved by the Ethics Committee of the Sixth Affiliated Hospital of Sun Yat-sen University (2021ZSLYEC-78), and registered at Clinicaltrials.gov (NCT04853147).
Sampling Method: Probability Sample
Enrollment: 1154 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Delayed clinically important postoperative nausea and vomiting | Every 24 hours after surgery (at 2-day, 3-day, 4-day and 5-day)
  A postoperative nausea and vomiting severity score of ≥ 5 based on the simplified postoperative nausea and vomiting impact scoring system, assessed between 25 and 120 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhinan Zheng, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Anesthesia, The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Nino MC, Calle S, Ruiz D, Baron MA, Cohen D, Martinez JE, Benitez DS, Mejia JA, Guerra JD, Kattah L. Rethinking postoperative nausea and vomiting prevention beyond perioperative medications. J Clin Anesth. 2024 Aug;95:111457. doi: 10.1016/j.jclinane.2024.111457. Epub 2024 Mar 29. No abstract available. PMID 38554569
- [Background] Chow R, Navari RM, Terry B, DeAngelis C, Prsic EH. Olanzapine 5 mg vs 10 mg for the prophylaxis of chemotherapy-induced nausea and vomiting: a network meta-analysis. Support Care Cancer. 2022 Feb;30(2):1015-1018. doi: 10.1007/s00520-021-06606-x. No abstract available. PMID 34613472
- [Background] White PF, Sacan O, Nuangchamnong N, Sun T, Eng MR. The relationship between patient risk factors and early versus late postoperative emetic symptoms. Anesth Analg. 2008 Aug;107(2):459-63. doi: 10.1213/ane.0b013e31817aa6e4. PMID 18633024
- [Background] Mraovic B, Simurina T. Effects of an intravenous lidocaine bolus before tracheal extubation on recovery after breast surgery - Lidocaine at the End (LATE) study: a randomized controlled clinical trial. Croat Med J. 2023 Aug 31;64(4):222-230. doi: 10.3325/cmj.2023.64.222. PMID 37654034
- [Background] Hermans V, De Pooter F, De Groote F, De Hert S, Van der Linden P. Effect of dexamethasone on nausea, vomiting, and pain in paediatric tonsillectomy. Br J Anaesth. 2012 Sep;109(3):427-31. doi: 10.1093/bja/aes249. PMID 22879656
- [Background] Gan TJ, Gu J, Singla N, Chung F, Pearman MH, Bergese SD, Habib AS, Candiotti KA, Mo Y, Huyck S, Creed MR, Cantillon M; Rolapitant Investigation Group. Rolapitant for the prevention of postoperative nausea and vomiting: a prospective, double-blinded, placebo-controlled randomized trial. Anesth Analg. 2011 Apr;112(4):804-12. doi: 10.1213/ANE.0b013e31820886c3. Epub 2011 Mar 8. PMID 21385988
- [Background] Mc Loughlin S, Terrasa SA, Ljungqvist O, Sanchez G, Garcia Fornari G, Alvarez AO. Nausea and vomiting in a colorectal ERAS program: Impact on nutritional recovery and the length of hospital stay. Clin Nutr ESPEN. 2019 Dec;34:73-80. doi: 10.1016/j.clnesp.2019.08.010. Epub 2019 Sep 11. PMID 31677715